CLINICAL TRIAL: NCT07399288
Title: Postherpetic Neuralgia After Herpes Zoster and Risk of Incident Dementia: Real-World Evidence From an International Matched Cohort With Landmark Analysis
Brief Title: Postherpetic Neuralgia After Herpes Zoster and Incident Dementia Risk
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH114-REC3-226
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Herpes Zoster; Dementia; Postherpetic Neuralgia (PHN)
Keywords: Landmark analysis; Propensity score matching; TriNetX; Alzheimer disease; Vascular dementia; Zoster vaccination; Negative control outcome
MeSH Terms: conditions — Herpes Zoster; Dementia; Neuralgia, Postherpetic; Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postherpetic neuralgia (PHN): Adults aged 40 to 120 years with incident herpes zoster between 1 October 2015 and 31 December 2024 who had a recorded postherpetic neuralgia diagnosis (ICD-10-CM B02.22 or B02.29) between 90 and 365 days after the index herpes zoster date. Follow-up begins at a 365-day landmark after index among individuals alive and free of dementia at the landmark.
  Interventions: Other: Exposure: postherpetic neuralgia
- Non-PHN comparator: Adults aged 40 to 120 years with incident herpes zoster between 1 October 2015 and 31 December 2024 with no recorded postherpetic neuralgia diagnosis (ICD-10-CM B02.22 or B02.29) within 365 days after the index herpes zoster date. Follow-up begins at a 365-day landmark after index among individuals alive and free of dementia at the landmark.

INTERVENTIONS:
Other: Exposure: postherpetic neuralgia — This is an observational study and no treatment is assigned by the investigators. The intervention of interest is exposure status defined by recorded diagnoses of postherpetic neuralgia after herpes zoster, based on ICD-10-CM codes B02.22 or B02.29 within 90 to 365 days after the index herpes zoster date.
  Groups: Postherpetic neuralgia (PHN)

SUMMARY:
This retrospective observational cohort study uses de-identified electronic health record data from the TriNetX Global Collaborative Network to evaluate whether postherpetic neuralgia after herpes zoster is associated with an increased risk of incident dementia. Adults aged 40 to 120 years with incident herpes zoster between 1 October 2015 and 31 December 2024 are identified using diagnostic codes. Postherpetic neuralgia is defined by International Classification of Diseases, 10th Revision, Clinical Modification (ICD-10-CM) codes B02.22 or B02.29 recorded between 90 and 365 days after the index herpes zoster date, and comparators have no such codes within 365 days after index. The primary analysis uses 1:1 propensity score matching and a 365-day landmark design, including only individuals alive and free of dementia at the landmark. Time-to-event analyses estimate hazard ratios for incident dementia and related outcomes.

DETAILED DESCRIPTION:
Data source and study design This is a retrospective cohort study using de-identified electronic health record data accessed through the TriNetX platform. The primary analysis is conducted in the TriNetX Global Collaborative Network. Replication is performed in the TriNetX Asia Pacific (APAC) network as a geographic validation.

Population and index date Eligible individuals are aged 40 to 120 years and have an incident herpes zoster diagnosis (ICD-10-CM B02) recorded between 1 October 2015 and 31 December 2024, with a 3-year washout period free of herpes zoster before the index date. Baseline covariates are assessed up to 1 day before the index date.

Exposure definition Postherpetic neuralgia is defined by ICD-10-CM codes B02.22 or B02.29 recorded between 90 and 365 days after the index date. The comparator cohort includes individuals with incident herpes zoster and no record of B02.22 or B02.29 within 365 days after the index date. A prespecified stricter exposure definition requires at least two postherpetic neuralgia codes separated by at least 30 days.

Landmark design and follow-up The primary analysis uses a 365-day landmark after the index date. Only individuals alive and free of the specified outcome at the landmark enter the risk set. Follow-up starts at the landmark and continues until the first record of the outcome, death, loss to follow-up, or 31 December 2024.

Matching and analysis Cohorts are matched 1:1 using nearest neighbour propensity score matching with a caliper of 0.1. Balance is assessed using standardised mean differences. Time-to-event analyses use Kaplan-Meier methods and Cox proportional hazards models, reporting hazard ratios with 95% confidence intervals.

Outcomes The primary outcome is incident all-cause dementia defined by ICD-10-CM codes F01, F02, F03, or G30. Prespecified secondary outcomes include Alzheimer disease, vascular dementia, other or unspecified dementia, all-cause mortality, ischaemic stroke, and hip fracture. The Benjamini-Hochberg false discovery rate is applied to the six secondary outcomes only. A negative control outcome of acute appendicitis (ICD-10-CM K35) is included to assess residual bias.

Sensitivity and validation analyses Prespecified analyses include an alternative 730-day landmark, the stricter postherpetic neuralgia definition, additional adjustment for recorded zoster vaccination as a baseline covariate, and replication in the TriNetX APAC network using prespecified matching settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 to 120 years with an incident herpes zoster diagnosis recorded between 1 October 2015 and 31 December 2024 in the TriNetX network.
* A 3-year washout period with no recorded herpes zoster diagnosis before the index date.
* Eligible for analysis at the 365-day landmark after the index date, defined as being alive and free of the specified outcome at the landmark.

Exclusion Criteria:

* Any record of the specified outcome before the 365-day landmark.
* Missing data elements required to define exposure status within the prespecified time window.

Ages: 40 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises adults aged 40 to 120 years with incident herpes zoster identified in the TriNetX Global Collaborative Network from 1 October 2015 to 31 December 2024. Exposure groups are defined by the presence or absence of recorded postherpetic neuralgia diagnoses within 90 to 365 days after the index herpes zoster date. Follow-up for outcomes starts at a 365-day landmark after index among individuals alive and free of the outcome at the landmark. Replication analyses are performed in the TriNetX Asia Pacific (APAC) network.
Sampling Method: Non-Probability Sample
Enrollment: 68786 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Incident all-cause dementia | From the 365-day landmark after the index herpes zoster date to the earliest of the first record of dementia, death, loss to follow-up, or 31 December 2024.
  Incident all-cause dementia is identified using ICD-10-CM codes F01, F02, F03, or G30. Individuals with any record of dementia before the 365-day landmark are excluded from the risk set.

SECONDARY OUTCOMES:
Alzheimer disease | From the 365-day landmark after the index herpes zoster date to the earliest of the first record of Alzheimer disease, death, loss to follow-up, or 31 December 2024.
  Incident Alzheimer disease is identified using ICD-10-CM code G30. Individuals with any record of Alzheimer disease before the 365-day landmark are excluded from the risk set.
Vascular dementia | From the 365-day landmark after the index herpes zoster date to the earliest of the first record of vascular dementia, death, loss to follow-up, or 31 December 2024.
  Incident vascular dementia is identified using ICD-10-CM code F01. Individuals with any record of vascular dementia before the 365-day landmark are excluded from the risk set.
Other or unspecified dementia | From the 365-day landmark after the index herpes zoster date to the earliest of the first record of other or unspecified dementia, death, loss to follow-up, or 31 December 2024.
  Incident other or unspecified dementia is identified using ICD-10-CM codes F02 or F03. Individuals with any record of these diagnoses before the 365-day landmark are excluded from the risk set.
All-cause mortality | From the 365-day landmark after the index herpes zoster date to the earliest of death, loss to follow-up, or 31 December 2024.
  All-cause mortality is identified using the death indicator available within the TriNetX network.
Ischaemic stroke | From the 365-day landmark after the index herpes zoster date to the earliest of the first record of ischaemic stroke, death, loss to follow-up, or 31 December 2024.
  Incident ischaemic stroke is identified using ICD-10-CM code I63. Individuals with any record of ischaemic stroke before the 365-day landmark are excluded from the risk set.
Hip fracture | From the 365-day landmark after the index herpes zoster date to the earliest of the first record of hip fracture, death, loss to follow-up, or 31 December 2024.
  Incident hip fracture is identified using ICD-10-CM codes S72.0, S72.1, or S72.2. Individuals with any record of hip fracture before the 365-day landmark are excluded from the risk set.

OTHER OUTCOMES:
Acute appendicitis (negative control outcome) | From the 365-day landmark after the index herpes zoster date to the earliest of the first record of acute appendicitis, death, loss to follow-up, or 31 December 2024.
  Incident acute appendicitis is identified using ICD-10-CM code K35. Individuals with any record of acute appendicitis before the 365-day landmark are excluded from the risk set.

CONTACTS AND LOCATIONS:
Overall Officials: En-Bo Wu, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taichung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) cannot be shared publicly because the TriNetX data are available only to subscribing organisations under licence agreements and governance controls. Investigators access de-identified records within the platform and are not permitted to download or redistribute line-level data. Researchers with access to TriNetX can reproduce the analysis using the cohort definitions and query parameters reported in the study.

REFERENCES:
- [Background] Stein E, Huser M, Amirian ES, Palchuk MB, Brown JS. TriNetX Dataworks-USA: Overview of a Multi-Purpose, De-Identified, Federated Electronic Health Record Real-World Data and Analytics Network and Comparison to the US Census. Pharmacoepidemiol Drug Saf. 2025 Sep;34(9):e70198. doi: 10.1002/pds.70198. PMID 40915660
- [Background] Warren-Gash C, Williamson E, Shiekh SI, Borjas-Howard J, Pearce N, Breuer JM, Smeeth L. No evidence that herpes zoster is associated with increased risk of dementia diagnosis. Ann Clin Transl Neurol. 2022 Mar;9(3):363-374. doi: 10.1002/acn3.51525. Epub 2022 Feb 16. PMID 35170873
- [Background] Forbes HJ, Thomas SL, Smeeth L, Clayton T, Farmer R, Bhaskaran K, Langan SM. A systematic review and meta-analysis of risk factors for postherpetic neuralgia. Pain. 2016 Jan;157(1):30-54. doi: 10.1097/j.pain.0000000000000307. PMID 26218719
- See also: TriNetX: Real-world data for the life sciences and healthcare — https://trinetx.com